CLINICAL TRIAL: NCT04814238
Title: Multicentre Registry of Minimally Invasive Aorta and Aortic Root Surgeries in Patients With Aortic Aneurysms
Brief Title: Minimally Invasive Aortic Root and Aorta surGery rEgistry
Acronym: MIRAGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nicolaus Copernicus University (Other)
Collaborators: Maastricht University Medical Center (Other); Prof. Franciszek Lukaszczyk Memorial Oncology Center (Other); Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Mariusz Kowalewski, MD, PhD, Nicolaus Copernicus University
Other Study IDs: #1/2021
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Aortic Aneurysm, Thoracic
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- mini-David
  Interventions: Procedure: Aortic Root Surgery
- mini-Yacoub
  Interventions: Procedure: Aortic Root Surgery
- mini-Bentall
  Interventions: Procedure: Aortic Root Surgery

INTERVENTIONS:
Procedure: Aortic Root Surgery — First time, isolated, minimally invasive (mini-sternotomy, RALT) aortic root or aorta surgery
  Other Names: Ascending Aorta Aneurysm Surgery, Aortoplasty, Supracoronary Replacement

SUMMARY:
Minimally invasive aortic valve (AV) surgery has become widely accepted alternative to standard sternotomy. Despite possible reduction in morbidity, this approach is not routinely performed for aortic surgery. Evidence exists, however, on safety of this approach together with promising results regarding its long-term durability. The MIRAGE Registry is aimed to collect and analyse the data from multiple aortic excellence centres and to analyse them in numerous clinical scenarios.

ELIGIBILITY:
Inclusion Criteria:

* isolated, first time aortic root or aorta surgery

Exclusion Criteria:

* active aortic valve endocarditis, redo surgery, acute type A dissection, and concomitant cardiac procedures.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients undergoing minimally-invasive aortic root and aorta surgery.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Early (in-hospital/30-day) mortality | 30 days

SECONDARY OUTCOMES:
Freedom from reoperation | 5 years
Long-term mortality | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Suwalski, MD, PhD, Study Director — Department of Cardiac Surgery, Central Clinical Hospital of the Ministry of Interior and Administration, Centre of Postgraduate Medical Education, Warsaw, Poland; Jakub Staromłyński, MD, PhD, Principal Investigator — Department of Cardiac Surgery, Central Clinical Hospital of the Ministry of Interior and Administration, Centre of Postgraduate Medical Education, Warsaw, Poland; Mariusz Kowalewski, MD, PhD, Principal Investigator — Department of Cardiac Surgery, Central Clinical Hospital of the Ministry of Interior and Administration, Centre of Postgraduate Medical Education, Warsaw, Poland
Locations (1):
- Department of Cardiac Surgery, Central Clinical Hospital of the Ministry of Interior and Administration, Centre of Postgraduate Medical Education, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Staromlynski J, Kowalewski M, Sarnowski W, Smoczynski R, Witkowska A, Bartczak M, Drobinski D, Wierzba W, Suwalski P. Midterm results of less invasive approach to ascending aorta and aortic root surgery. J Thorac Dis. 2020 Nov;12(11):6446-6457. doi: 10.21037/jtd-20-2165. PMID 33282347
- [Background] Staromlynski J, Kowalewski M, Smoczynski R, Suwalski P. Minimally invasive approach to ascending aorta and aortic root surgery. Interact Cardiovasc Thorac Surg. 2021 Jan 1;32(1):163. doi: 10.1093/icvts/ivaa214. No abstract available. PMID 33372227